CLINICAL TRIAL: NCT04902612
Title: Prospective, Controlled, Randomized, Double-blind, Premarket Multi-centre Study on the Performance of HM242-Solution vs Comparator in Patients Under Condition of Venous Leg Ulcer
Brief Title: HM242-Solution vs Comparator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPM-G-H-2003
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM242-Solution (Experimental)
  Interventions: Device: HM242-Solution
- Saline (Active Comparator)
  Interventions: Device: Saline

INTERVENTIONS:
Device: HM242-Solution — HM242-Solution compared to Saline compared in patients with a venous leg ulcer
  Arms: HM242-Solution
Device: Saline — HM242-Solution compared to Saline compared in patients with a venous leg ulcer
  Arms: Saline

SUMMARY:
The objectives of this study include investigating the performance of HM242-Solution compared to normal Saline with respect to venous leg ulcer healing. Saline is widely used for venous leg ulcer cleansing and has served as comparator or standard treatment in clinical trials evaluating new cleansing products to prove that it is as good as the standard treatment. Data will also be collected on the patients' quality of life and any adverse events that may arise during the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of at least 18 years at the time of enrolment
* Has the legal capacity and is able to understand the nature, risks, significance and scope of the clinical trial and to determine his or her will accordingly
* Signed form of consent, including the understanding of and willingness by the patient to participate in the clinical study and ability to comply with study procedures and study visit schedule
* Patients must be willing to have all dressing changes performed by the wound specialist, with no treatments at home
* Presence of at least one venous ulcer of the lower leg extending through the full thickness of the skin but not down to muscle, tendon or bone
* Size of study ulcer ≥ 2cm² and ≤ 100cm² measured using the tracing method
* Presence of venous leg ulcer for at least 6 weeks, but not longer than 12 months
* Ankle Brachial Pressure Index (ABI) > 0.75
* In the case of a female patient of childbearing potential, willingness to use highly effective methods of contraception (failure rate of < 1% when used consistently and correctly); acceptable contraceptive measures in this trial are: combined pill and progestin-only pill, contraceptive patch, ring or injection, Etonogestrel implant, intrauterine device (IUD) (copper and Levonogestrel), male sterilization (vasectomy), female sterilization (abdominal, laparoscopic, hysteroscopic), or sexual abstinence.

Exclusion Criteria:

* Patients kept in an institution due to an official or court order
* Patients dependent on the Sponsor, Investigator or Site
* Patients suspected of having SARS-CoV-2 infection or COVID-19 disease
* Study ulcer judged by the Investigator to be caused by a medical condition other than venous insufficiency
* Study ulcer with signs and symptoms of infection, or under suspicion of cancer
* Study ulcer under treatment with topical antimicrobials within past two weeks or systemic antimicrobial treatment within past two weeks
* More than two venous leg ulcers or more than two chronic wounds
* Dementia stage greater than 3 according to Reisberg
* Known allergies against wound dressings used in the study
* Known chronical skin diseases, dermatoses, or known allergies or other conditions which might trigger dermatitis
* Acute cases of substance use disorders (ICD-10 F1x.1 or F1x.2)
* Buerger's disease
* Participation in Medical Device trials less than 4 weeks ago or participation in Drug trials less than six months ago
* Terminally ill patients
* Patients with poorly managed diabetes mellitus: absence of a glycated hemoglobin test within the last 3 months or a result of HbA1c ≥ 8% not older than 3 months, or a major diabetes-related incident within the past 4 weeks
* Ulcers of diabetic origin
* Patients under treatment with systemic corticosteroids, immunosuppressants, cytotoxic chemotherapy, or radiotherapy
* Presence of one or more medical conditions (other than venous insufficiency and diabetes) as determined by medical history, which:
* Is known to interfere with the wound healing process (e.g. arteriopathy, vasculitis, rheumatoid arthritis, systemic lupus erythematosus, other auto-immune diseases, cancer, immunodeficiency, severe lymphedema of the leg, thrombophilia)
* In the opinion of the Investigator, would make the patient an inappropriate candidate for this venous ulcer healing study (e.g. malnutrition, hygiene, obesity)
* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to demonstrate that the HM242-Solution performs at least comparably to Saline regarding wound healing. | 28 days
  The primary variable is defined as the relative reduction of the wound area of a patient in percentage 28 days (4 weeks) after baseline. The wound size area is measured on site by the Tracing method.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Asl Napoli 3 Sud, Gragnano, Napoli
  - Dept. of Clinical and Experimental Medicine University of Pisa, Pisa, Toscany

IPD SHARING:
Plan to Share IPD: No